CLINICAL TRIAL: NCT04585230
Title: Prospective Blinded Randomized Controlled Trial Evaluating the Outcomes of Cannabinoid (CBD) Roll-on Topical Stick in Primary Total Knee Arthroplasty
Brief Title: A Study to Evaluate the Outcomes of Cannabinoid (CBD) Roll-on Topical Stick in Primary Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JLON20P.202
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pain, Joint; Pain, Postoperative; Total Knee Arthroplasty
MeSH Terms: conditions — Arthralgia; Pain, Postoperative | interventions — Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: (CBD + MO cohort) (Active Comparator): Roll on stick containing CBD and mineral oils (CBD + MO cohort)
  Interventions: Drug: CBD; Drug: Mineral Oil
- Group 2: (MO cohort) (Active Comparator): Roll on stick containing mineral oils only (MO cohort)
  Interventions: Drug: Mineral Oil
- Group 3: (CBD Cohort) (Active Comparator): Roll on stick containing CBD only (CBD cohort)
  Interventions: Drug: CBD
- Group 4: (Roll-on stick only with NO CBD or MO-placebo cohort) (Placebo Comparator): Roll on stick with neither CBD nor essential oils (Roll-on stick only with NO CBD or MO-placebo cohort)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD — CBD oil Roll-On Stick
  Arms: Group 1: (CBD + MO cohort); Group 3: (CBD Cohort)
Drug: Mineral Oil — Mineral Oil- Roll on Stick
  Arms: Group 1: (CBD + MO cohort); Group 2: (MO cohort)
Drug: Placebo — Roll- On stick with no CBD and no Mineral Oil
  Arms: Group 4: (Roll-on stick only with NO CBD or MO-placebo cohort)

SUMMARY:
Total knee arthroplasty (TKA) is one the most common surgical treatments performed for end stage degenerative arthritis of the knee. More than 700,000 procedures are currently performed yearly in the United States. This procedure usually results in moderate-to-severe pain in the immediate post-operative period. Optimal pain control may allow early mobilization, accelerate rehabilitation, improve patient satisfaction, decrease length-of-stay, and optimize functional outcomes. The challenge, however, is to manage pain with alternative methods, reducing the role of opiate medications, which are highly addictive with myriad side effects.

In this prospective randomized double-blinded controlled study, the investigators aim to evaluate the benefits of an over-the-counter (OTC) transdermal CBD preparation in patients undergoing primary total knee arthroplasty as a novel adjunct to the standard multi-modal analgesic regimen, to reduce postoperative pain and reduce the need for opiates after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have general anesthesia
2. Patients who have documented allergic reactions to ropivacaine in the local infiltration agents
3. Patients who have a contra-indication to the use of non-steroidal anti-inflammatory medications or are using therapeutic anticoagulation precluding them from using non-steroidal anti-inflammatory medications
4. Patients unable to complete a 100-ft walk baseline
5. Patients undergoing total knee arthroplasty as a conversion procedure following previous surgery
6. Patients undergoing TKA for posttraumatic arthritis
7. Patients undergoing TKA for steroid-induced or spontaneous avascular necrosis
8. Workers compensation patients
9. Patients refusing or not candidates for peripheral nerve blocks
10. Patients undergoing unicompartmental knee arthroplasty
11. Patients undergoing patellofemoral arthroplasty
12. Patients undergoing bilateral simultaneous or sequential primary total knee arthroplasty within the same hospital stay
13. Patients who have previously reported allergy to tetrahydrocannabinol or other cannabinoid compounds or develop allergic reactions to the formulation following use
14. Patients who are pregnant or choosing to be pregnant during the 6-week study period or are breast feeding during the study period
15. Patients who are on chronic narcotics pre-operatively
16. Patients who have end-stage cirrhosis, end-stage renal failures, or psychiatric conditions preventing adequate assessment of study outcome metrics
17. Patients with adequate cognitive function to participate and complete questionnaires for the study.
18. Patients unable or unwilling to follow-up and complete questionnaires for the study
19. Patients with active cancer and undergoing treatment precluding the assessment of outcome metrics
20. Patients with a history or diagnosis of chronic pain syndrome or Complex regional pain syndrome (CRPS)
21. Patients who are determined to be in severe pain from other concomitant conditions

Exclusion Criteria:

1. patients <18 and >80
2. any patient who does not meet the inclusion criteria listed for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-10-12 (Estimated); Primary Completion 2021-05-28 (Estimated); Study Completion 2021-05-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative change in pain and change the need for opiates after total knee arthroplasty. | 14 days
  opioid consumption after surgery will be calculated in morphine equivalents

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States